CLINICAL TRIAL: NCT00193492
Title: Rituximab +/- Bevacizumab in the Treatment of Patients With Follicular Non-Hodgkin's Lymphoma: A Randomized, Phase II Trial
Brief Title: A Study of Rituximab and Bevacizumab in Patients With Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 37; U3234s (Other: Genentech-Roche)
Record Dates: First submitted 2005-08-22; First posted 2005-09-19 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Lymphoma, Follicular
Keywords: Lymphoma; Bevacizumab; Rituximab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — Bevacizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Active Comparator): All patients will receive rituximab 375mg/m2 administered by slow IV infusion weekly for 4 consecutive weeks (days 1, 8, 15, and 22). Patients who have objective response or stable disease at week 12 reevaluation will receive 4 additional doses of rituximab (375 mg/m2) administered in months 3 (week 12), 5, 7, and 9.
  Interventions: Drug: Rituximab
- Rituximab/Bevacizumab (Experimental): All patients will receive rituximab 375mg/m2 administered by slow IV infusion weekly for 4 consecutive weeks (days 1, 8, 15, and 22). During the 4-week course of rituximab, all patients will receive 2 doses of bevacizumab 10mg/kg IV, given on Days 3 and 15. The first dose will be given on Day 3, following rituximab on Day 1. If both drugs are well tolerated during the first dose, rituximab and bevacizumab should be given on the same day for the Day 15 dose and all subsequent doses.
  Interventions: Drug: Bevacizumab; Drug: Rituximab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Rituximab/Bevacizumab
Drug: Rituximab
  Other Names: Rituxan; MabThera

SUMMARY:
The purpose of this study is to assess the feasibility, efficacy and safety of adding bevacizumab to rituximab compared to rituximab alone in patients with previously treated follicular non-hodgkin's lymphoma (NHL) whose disease has progressed following at least one previous chemotherapy regimen and not more than 2 previous chemotherapy regimens.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will randomly be assigned to one of two treatment arms:

* Rituximab
* Rituximab + bevacizumab

For every 2 patients randomized, 1 will receive treatment number 1 (rituximab), and 1 patient will receive treatment number 2 (rituximab + bevacizumab). This is not a blinded study, so both the patient and doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, you must meet the following criteria:

* Follicular NHL, grades 1 or 2 confirmed by a biopsy sample
* 18 years of age or older
* Evidence of disease progression at time of study entry
* Must have had at least one previous chemotherapy regimen and not more than two previous chemotherapy regimens.
* Patients who have received previous rituximab are eligible as long as progression occurred more than six months following completion of previous rituximab therapy.
* Measurable or evaluable disease
* Able to perform activities of daily living without considerable assistance
* Adequate bone marrow, kidney, and liver function
* Signed informed consent obtained prior to initiation of any study-specific procedures or treatment.

Exclusion Criteria:

You cannot participate in the study if any of the following apply to you:

* Treatment with more than two previous chemotherapy regimens
* Prior treatment with bevacizumab or other similar agents
* Progressive NHL less than 6 months after receiving previous rituximab
* More than 1 prior treatment with investigational agents within 4 weeks prior to entering this study
* Spread of NHL to brain or nervous system
* History of any other uncontrolled or significant disease or medical condition that may put them at high risk for treatment complications with these agents

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (22):
- United States (22):
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Watson Clinic for Cancer Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Baptist Hospital East, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Berks Hematology Oncology Associates, West Reading, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: All patients will receive rituximab 375mg/m2 administered by slow IV infusion weekly for 4 consecutive weeks (days 1, 8, 15, and 22). Patients who have objective response or stable disease at week 12 reevaluation will receive 4 additional doses of rituximab (375 mg/m2) administered in months 3 (week 12), 5, 7, and 9.
  Rituximab
- Rituximab/Bevacizumab: All patients will receive rituximab 375mg/m2 administered by slow IV infusion weekly for 4 consecutive weeks (days 1, 8, 15, and 22). During the 4-week course of rituximab, all patients will receive 2 doses of bevacizumab 10mg/kg IV, given on Days 3 and 15. The first dose will be given on Day 3, following rituximab on Day 1. If both drugs are well tolerated during the first dose, rituximab and bevacizumab should be given on the same day for the Day 15 dose and all subsequent doses.
  Bevacizumab
  Rituximab
Period: Overall Study
Arm/Group | Rituximab | Rituximab/Bevacizumab
Started | 31 | 29
Completed | 14 | 14
Not Completed | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Rituximab/Bevacizumab | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Median (Full Range); unit: years] | 65 [47 to 80] | 68 [45 to 91] | 67 [45 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 18 | 13 | 31
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab | Rituximab/Bevacizumab
Number analyzed (Participants) | 31 | 29
percentage of participants | 42 [25 to 61] | 48 [29 to 67]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death or Disease Progression from NHL. Progression is defined using International Workshop Response Criteria for Non-Hodgkin's Lymphoma as - enlargment of liver/spleen, new sites, new or increased malignancy in lymph nodes, new or increased lymph node masses or reappearance of disease in bone marrow.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab | Rituximab/Bevacizumab
Number analyzed (Participants) | 31 | 29
months | 10.4 [4.4 to 15.9] | 20.7 [13.8 to 54.4]

ADVERSE EVENTS:
Arm/Group | Rituximab | Rituximab/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/31 | 8/29
Other Adverse Events (participants affected / at risk) | 29/31 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=31) | Rituximab/Bevacizumab (N=29)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Psychiatric disorders - Other, dementia (Psychiatric disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Rectal Perforation (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=31) | Rituximab/Bevacizumab (N=29)
Fatigue (General disorders) | 17 | 20
Pain (General disorders) | 14 | 17
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 10
White blood cell decreased (Investigations) | 6 | 13
Anemia (Blood and lymphatic system disorders) | 11 | 7
Platelet count decreased (Investigations) | 8 | 8
Hypertension (Vascular disorders) | 3 | 12
Nausea (Gastrointestinal disorders) | 6 | 9
Headache (Nervous system disorders) | 3 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 11
Proteinuria (Renal and urinary disorders) | 1 | 11
Allergic reaction (Immune system disorders) | 8 | 2
Infections and infestations - Other (Infections and infestations) | 3 | 7
Edema (General disorders) | 7 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 5
Neutrophil count decreased (Investigations) | 4 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 6
Insomnia (Psychiatric disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 3 | 3
Dizziness (Nervous system disorders) | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 5
Alkaline phosphatase increased (Investigations) | 2 | 3
Blood and lymphatic system disorders - Other, hematocrit decreased (Blood and lymphatic system disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Fever (General disorders) | 3 | 2
Metabolism and nutrition disorders - Other, hyperchloremia (Metabolism and nutrition disorders) | 1 | 4
Psychiatric disorders - Other, mood alteration NOS (Psychiatric disorders) | 1 | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3
Chills (General disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Creatinine increased (Investigations) | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
General disorders and administration site conditions - Other, hemorrhage (General disorders) | 0 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2
Lymphocyte count decreased (Investigations) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Rhinitis infective (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Urinary frequency (Renal and urinary disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the propsed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites